CLINICAL TRIAL: NCT06297668
Title: A Phase I, Randomized, Partial Double-blind, Single-dose, 3-Way Cross-over Study to Assess the Total Systemic Exposure of Budesonide, Glycopyrronium, and Formoterol for BGF MDI HFO Compared With BGF MDI HFA Using an AeroChamber Plus Flow-Vu Spacer and to Compare the Total Systemic Exposure of BGF MDI HFO With a Spacer to BGF MDI HFO Without a Spacer
Brief Title: A Study to Assess the Pharmacokinetics and Safety of Budesonide, Glycopyrronium, & Formoterol (BGF) Metered Dose Inhaler (MDI) With a Next-Generation Propellant (NGP) With a Spacer, BGF MDI Hydrofluoroalkane (HFA) With a Spacer, as Well as BGF MDI NGP Without a Spacer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Collaborators: Parexel (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: D5985C00008; 2023-504089-43-00 (Registry Identifier: CTIS)
Record Dates: First submitted 2024-03-01; First posted 2024-03-07 (Actual); Last update posted 2025-08-13 (Actual); Status verified 2025-08

CONDITIONS: Chronic Obstructive Pulmonary Disease
Keywords: Metered Dose Inhalers (MDI); Propellant; Next Generation Propellant (NGP); Inhaled Corticosteroid (ICS); Long-acting muscarinic antagonist (LAMA); Long-acting beta2 agonist (LABA); Total Systemic exposure; Healthy participants
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: Yes

ARMS (3):
- BGF MDI HFA (Active Comparator): Budesonide/Glycoperronium/formoterol fumarate pressurised inhalation suspension 160/7.2/4.8 μg per actuation, hydroﬂuoroalkane with AeroChamber Plus Flow-Vu spacer-reference formulation
  Interventions: Drug: Treatment A: BGF MDI HFA; Device: AeroChamber Plus Flow-Vu spacer
- BGF MDI HFO with spacer (Active Comparator): Budesonide/Glycoperronium/formoterol fumarate pressurised inhalation suspension 160/7.2/4.8 μg per actuation, hydrofluoroolefin with AeroChamber Plus Flow-Vu spacer-test formulation
  Interventions: Drug: Treatment B: BGF MDI HFO; Device: AeroChamber Plus Flow-Vu spacer
- BGF MDI HFO without spacer (Active Comparator): Budesonide/Glycoperronium/formoterol fumarate pressurised inhalation suspension 160/7.2/4.8 μg per actuation, hydrofluoroolefin without AeroChamber Plus Flow-Vu spacer
  Interventions: Drug: Treatment C: BGF MDI HFO

INTERVENTIONS:
Drug: Treatment A: BGF MDI HFA — Participants will receive 4 inhalations of BGF MDI HFA as a single dose with AeroChamber Plus Flow-Vu spacer.
  Arms: BGF MDI HFA
Drug: Treatment B: BGF MDI HFO — Participants will receive 4 inhalations of BGF MDI HFO as a single dose with AeroChamber Plus Flow-Vu spacer.
  Arms: BGF MDI HFO with spacer
Drug: Treatment C: BGF MDI HFO — Participants will receive 4 inhalations of BGF MDI HFO as a single dose without spacer.
  Arms: BGF MDI HFO without spacer
Device: AeroChamber Plus Flow-Vu spacer — Participants will receive 4 inhalations of BGF MDI HFA (Treatment A) and BGF MDI HFO (Treatment B) as a single dose with spacer.
  Arms: BGF MDI HFA; BGF MDI HFO with spacer

SUMMARY:
This study aims to assess the effect on total systemic exposure and to characterize exposure BGF MDI HFO with a spacer compared to without a spacer; also, to demonstrate that total systemic exposure of BGF when administered as MDI HFO with a spacer is not greater than BGF MDI HFA with a spacer.

DETAILED DESCRIPTION:
This is a Phase I, randomized, partial double-blind, single dose, three way cross-over study to assess the effect of total systemic exposure of BGF when administered as BGF MDI HFO compared with BGF MDI HFA Using an AeroChamber Plus Flow-Vu Spacer and to compare the Total Systemic Exposure of BGF MDI HFO with a Spacer to BGF MDI HFO without a Spacer in healthy participants (male or female).

The study will comprise of:

* A Screening Period of up to 27 days prior to first dosing.
* Three treatment periods: participants will be resident at the Clinical Unit from Day -1 until 24 hours after dosing with the final treatment, with a washout period of 3 to 7 days between each dose administration.
* Follow-up: a final Follow-up Phone Call within 5 to 7 days after the last administration of BGF MDI in Treatment Period 3.

Participants will receive all 3 treatments as a single dose (4 inhalations) (Treatment A [BGF MDI HFA with AeroChamber Plus Flow-Vu spacer - reference formulation], Treatment B [BGF MDI HFO with AeroChamber Plus Flow-Vu spacer - test formulation], and Treatment C [BGF MDI HFO without spacer]) (1 treatment per treatment period) in one of 6 possible treatment sequences; ABC, ACB, BAC, BCA, CAB, or CBA.

ELIGIBILITY:
Inclusion Criteria:

* Females must have a negative pregnancy test at screening and on admission to the Clinical Unit, must not be lactating, confirmed at screening.
* Women of childbearing potential who are sexually active with a non-sterilized male partner, must use 1 highly effective form of birth control from enrolment throughout the study and until at least 14 days after last dose of IMP. Women should be stable on their chosen method of birth control for at least 1 month from enrolment.
* Have a body mass index between 18 and 30 kg/m2 inclusive and weigh at least 50 kg.
* Have a Forced expiratory volume in the first second (FEV1) ≥ 80% of the predicted normal value and an FEV1/forced vital capacity> 70% regarding age, height, and ethnicity at screening.
* Demonstrate basic understanding of how to use an MDI device with and without a spacer after receiving training.
* Participants should be fully/sufficiently vaccinated as per local definitions against SARS-CoV-2 (in combination with confirmed past infections with SARS-CoV-2).

Exclusion Criteria:

* History or current evidence of any clinically significant disease or disorder, including endocrinological diseases, such as thyrotoxicosis, which, in the opinion of the investigator, may either put the participant at risk because of participation in the study, or influence the results through participation in the study.
* Participants who have previously received BGF MDI HFO.
* History of severe allergy/hypersensitivity or ongoing allergy/hypersensitivity, as judged by the investigator, or history of hypersensitivity to drugs with a similar chemical structure or class to BGF or to its excipients, such as norflurane.
* History or presence of gastrointestinal, hepatic, or renal disease, or any other condition known to interfere with absorption, distribution, metabolism, or excretion of drugs.
* Any clinically significant illness, medical/surgical procedure, or trauma within 4 weeks of the first administration of investigational medicinal product (IMP).
* History of narrow angle glaucoma or change in vision that may be relevant.
* History of symptomatic prostatic hypertrophy or bladder neck obstruction/urinary retention that, which in the opinion of the investigator, is clinically significant.
* Unresectable cancer that has not been in complete remission for at least 5 years.
* Any clinically significant abnormalities in clinical chemistry, hematology, or urinalysis results, at screening as judged by the investigator.
* Any clinically significant abnormal findings in physical examination or vital signs at screening, as judged by the investigator.
* Any clinically significant abnormalities on 12-lead ECG at screening, as judged by the investigator.
* Any positive result on screening for serum hepatitis B surface antigen or anti-hepatitis B core antibody, indicative of hepatitis B, hepatitis C antibody, or human immunodeficiency virus.
* Positive reverse transcription polymerase chain reaction test for SARS-CoV-2 prior to randomization.
* Participant has clinical signs and symptoms consistent with COVID-19, eg, fever, dry cough, dyspnea, sore throat, fatigue, new smell or taste disorder or confirmed infection by appropriate laboratory test within the last 4 weeks prior to screening or on admission.
* Participant who had severe course of COVID-19 (ie, hospitalization, extracorporeal membrane oxygenation, or mechanically ventilated).
* Recent (within 14 days prior to admission to the Clinical Unit) exposure to someone who has COVID-19 symptoms or tested positive for SARS-CoV-2.
* History of any respiratory disorders such as asthma, COPD, or idiopathic pulmonary fibrosis.
* Known or suspected history of drug abuse.
* Current smokers or those who have smoked or used nicotine products (including e-cigarettes) within the 3 months prior to screening.
* Use of drugs with enzyme-inducing properties such as St John's Wort within 3 weeks prior to the first administration of IMP.
* Use of any prescribed or non-prescribed medication including antacids, analgesics (other than paracetamol/acetaminophen), herbal remedies, megadose vitamins (intake of 20 to 600 times the recommended daily dose) and minerals during the 2 weeks prior to the first administration of IMP or longer if the medication has a long half-life.
* Known or suspected history of alcohol or drug abuse or excessive intake of alcohol.
* Excessive intake of caffeine-containing drinks or food (eg, coffee, tea, chocolate).

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 42 (Actual)
Dates: Start 2024-04-29 (Actual); Primary Completion 2024-06-11 (Actual); Study Completion 2024-06-11 (Actual)

PRIMARY OUTCOMES:
Area Under the Plasma Concentration-curve from Zero to the Last Quantifiable Concentration (AUClast) of BGF MDI | Day 1 and Day 2 of each treatment period (each treatment period is of 2 days)
  To assess that the total systemic exposure of budesonide, glycopyrronium, and formoterol administered as BGF MDI HFO with AeroChamber Plus Flow-Vu spacer does not exceed that with BGF MDI HFA with AeroChamber Plus Flow-Vu spacer.
Maximum Observed Concentration (Cmax) of BGF MDI | Day 1 and Day 2 of each treatment period (each treatment period is of 2 days)
  To assess that the total systemic exposure of budesonide, glycopyrronium, and formoterol administered as BGF MDI HFO with AeroChamber Plus Flow-Vu spacer does not exceed that with BGF MDI HFA with AeroChamber Plus Flow-Vu spacer.

SECONDARY OUTCOMES:
Area Under the Plasma Concentration-curve from Zero to the Last Quantifiable Concentration (AUClast) | Day 1 and Day 2 of each treatment period (each treatment period is of 2 days)
  To assess the relative bioavailability of budesonide, glycopyrronium, and formoterol administered as BGF MDI HFO with a spacer versus BGF MDI HFO without a spacer.
Maximum Observed Concentration (Cmax) | Day 1 and Day 2 of each treatment period (each treatment period is of 2 days)
  To assess the relative bioavailability of budesonide, glycopyrronium, and formoterol administered as BGF MDI HFO with a spacer versus BGF MDI HFO without a spacer.
Area Under the Plasma Concentration-time Curve From Time Zero to Infinity (AUCinf) | Day 1 and Day 2 of each treatment period (each treatment period is of 2 days)
  To characterize the PK parameters of budesonide, glycopyrronium, and formoterol administered as BGF MDI HFO (with and without spacer) and BGF MDI HFA with a spacer.
Time to Reach Maximum Observed Concentration (tmax) | Day 1 and Day 2 of each treatment period (each treatment period is of 2 days)
  To characterize the PK parameters of budesonide, glycopyrronium, and formoterol administered as BGF MDI HFO (with and without spacer) and BGF MDI HFA with a spacer.
Terminal Rate Constant (λz) | Day 1 and Day 2 of each treatment period (each treatment period is of 2 days)
  To characterize the PK parameters of budesonide, glycopyrronium, and formoterol administered as BGF MDI HFO (with and without spacer) and BGF MDI HFA with a spacer.
Half-life Associated with Terminal Slope (λz) of a Semi-logarithmic Concentration-time Curve (t1/2λz) | Day 1 and Day 2 of each treatment period (each treatment period is of 2 days)
  To characterize the PK parameters of budesonide, glycopyrronium, and formoterol administered as BGF MDI HFO (with and without spacer) and BGF MDI HFA with a spacer.
Mean Residence Time of the Unchanged Drug in the Systemic Circulation from Zero to Infinity (MRTinf) | Day 1 and Day 2 of each treatment period (each treatment period is of 2 days)
  To characterize the PK parameters of budesonide, glycopyrronium, and formoterol administered as BGF MDI HFO (with and without spacer) and BGF MDI HFA with a spacer.
Apparent Total Body Clearance of Drug from Plasma After Extravascular Administration (CL/F) | Day 1 and Day 2 of each treatment period (each treatment period is of 2 days)
  To characterize the PK parameters of budesonide, glycopyrronium, and formoterol administered as BGF MDI HFO (with and without spacer) and BGF MDI HFA with a spacer.
Apparent Volume of Distribution at Steady State Following Extravascular Administration (Vz/F) | Day 1 and Day 2 of each treatment period (each treatment period is of 2 days)
  To characterize the PK parameters of budesonide, glycopyrronium, and formoterol administered as BGF MDI HFO (with and without spacer) and BGF MDI HFA with a spacer.
Number of Participants with Adverse Events | From Baseline up to 48 days
  To assess the safety and tolerability of single doses of BGF MDI HFO (with and without spacer) and BGF MDI HFA with a spacer, in healthy participants.

CONTACTS AND LOCATIONS:
Locations (1):
- Research Site, Berlin, Germany

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers can request access to anonymized individual patient-level data from AstraZeneca group of companies sponsored clinical trials via the request portal Vivli.org. All requests will be evaluated as per the AZ disclosure commitment: https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure."Yes", indicates that AZ are accepting requests for IPD, but this does not mean all requests will be approved.
Time Frame: AstraZeneca will meet or exceed data availability as per the commitments made to the EFPIA/PhRMA Data-Sharing Principles. For details of our timelines, please refer to our disclosure commitment at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
Access Criteria: When a request has been approved AstraZeneca will provide access to the anonymized individual patient-level data via secure research environmentVivli.org. A Signed Data Usage Agreement (non-negotiable contract for data accessors) must be in place before accessing requested information.
URL: https://vivli.org/

REFERENCES:
- See also: CSR Synopsis — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217111&parentIdentifier=D5985C00008&attachmentIdentifier=a5202bd4-4afc-4ca6-879d-79e88a928efa&fileName=(278529)_D5985C00008_CSR_Synopsis_Final_Approved-Redacted.pdf&versionIdentifier=